CLINICAL TRIAL: NCT04666571
Title: Personalised Against Standard High Tibial Osteotomy, a Prospective Multi-centre Randomised Controlled Trial
Brief Title: Personalised Against Standard High Tibial Osteotomy
Acronym: PASHiOn
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Oxford (Other); 3D Metal Printing Ltd (Industry); Versus Arthritis (Other)
Responsible Party: Principal Investigator, Richie Gill, Professor of Healthcare Engineering, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCTRU263
Record Dates: First submitted 2020-11-26; First posted 2020-12-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Medial Knee Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised (TOKA) (Experimental): During HTO surgery, the personalised plate will be inserted below the knee.
  The investigational device and comparator are two types of metal plate used to fix the bone in place during a high tibial osteotomy (HTO).
  Interventions: Device: TOKA
- Standard (Tomofix or ActivMotion) (Active Comparator): During HTO surgery, the standard plate will be inserted below the knee.
  Interventions: Device: Tomofix or ActivMotion

INTERVENTIONS:
Device: TOKA — The device is a digitally planned (using individual CT scan measured anatomic data) personalised opening wedge high tibial osteotomy (HTO) procedure using a custom 3D printed surgical guide and plate.
  Other Names: Tailored Osteotomy Knee Alignment; Personalised HTO
  Arms: Personalised (TOKA)
Device: Tomofix or ActivMotion — The comparators, Tomofix and ActivMotion, are the most widely used devices for HTO procedures in the UK. Surgical procedures using the Tomofix and ActiveMotion are similar to TOKA, however, they are not patient specific and do not use custom-made plates.
  Other Names: Standard HTO; Generic HTO
  Arms: Standard (Tomofix or ActivMotion)

SUMMARY:
A study to compare the accuracy of achieving the planned correction between personalised (TOKA) high tibial osteotomy (HTO) procedure and standard generic HTO procedure.

DETAILED DESCRIPTION:
The trial design is a multi-centre, blinded, superiority two arm, parallel group design randomised controlled trial (RCT) of personalised (TOKA) versus standard high tibial osteotomy (HTO).

The aim of the PASHiOn trial is to establish whether digitally planned personalised HTO surgery (TOKA) increases the accuracy of bone correction in comparison to conventional HTO surgery. Embedded within the trial is a non-randomised pre-RCT technology check and safety assessment of 5 patients (Phase 1), followed by a randomised controlled trial of 88 (revised to 50) patients (Phase 2) .

During Phase 1 of the clinical investigation, 5 patients fulfilling the inclusion criteria will be recruited and assessed in an identical way to the 88 (revised to 50) patients recruited in the main trial, but without randomisation. Recruitment of the remaining patients (Phase 2) will take place after the six-week assessment on the fifth patient is complete and the oversight committee supports progression to Phase 2.

Patients will be randomised to Phase 2 in a 1:1 ratio and patients will be blinded as to which treatment arm they receive.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing High Tibial Osteotomy
* Male or Female, aged 18 to 65 years
* Primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD)
* Predominately diagnosed with unicompartmental medial osteoarthritis of the knee with the normal clinically acceptable level of other compartmental involvement
* Varus deformity <20 °
* BMI ≤ 35. An exemption to this may be made if the participant (in the investigators opinion) is suitable for surgery.
* Participant is willing and able to give informed consent for participation in the study.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Prisoners
* Participants with a known deep tissue sensitivity to device materials
* Participants with an active or suspected latent infection in or about the affected knee joint
* Participants who have received any orthopaedic surgical intervention to the lower extremities (excluding investigative surgery) within the past 12 months, or is expected to require any orthopaedic surgical intervention to the lower extremities, other than the HTO to be enrolled in this study, within the next 12 months (including intra-articular procedures).
* Participants who require bilateral HTO with surgery planned on their second knee within 6 months of their first operation (bilateral HTO patients are otherwise included).
* Participants who require bilateral HTO who have had a previous unsuccessful contralateral partial replacement or HTO
* Chronic heart failure (NYHA Stage ≥ 2)
* Neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device
* Systemic disease diagnosis (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's disease) leading to progressive bone deterioration.
* Participant is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* Participant is a smoker.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - To assess the safety of the TOKA device by determining the incidence/rate of Adverse Events, Adverse Device Effects, Serious Adverse Device Effects, Serious Adverse Events, Unexpected Serious Adverse Device Effects and complications. | 6 weeks post-surgery
  Incidence/rate of safety events - Adverse Events (AE), Adverse Device Effects (ADE), Serious Adverse Device Effects (SADEs), Serious Adverse Events (SAEs), Unexpected Serious Adverse Device Effects (SADEs) and complications.
Phase 2 - To establish if digitally planned personalised HTO surgery (TOKA) increases the accuracy of bone correction in comparison to conventional HTO surgery. | 9 months post-randomisation (6 months post-surgery)
  The absolute difference between planned and achieved coronal plane correction in terms of the hip-knee-ankle angle, (as measured from full length weight bearing x-rays)

SECONDARY OUTCOMES:
Number of patients (%) achieving a pre-specified difference between planned and achieved coronal plane correction | 9 months post-randomisation (6 months post-surgery)
  The number of patients who have difference between planned and achieved correction of less than 3 degrees in each treatment arm will be compared at 9 months post randomisation.
Change in coronal plane location of peak loading during gait, in comparison to baseline, measured by Video Vector | 9 months post-randomisation (6 months post-surgery)
  Video Vector Analysis (VVA) will be used at baseline and at 9 months post randomisation. VVA simultaneously records ground reaction force data from a force plate and video data from a video camera focussed on the lower limb of a participant. This enables the magnitude, orientation, and location of the ground reaction force to be determined relative to the limb under investigation.
Operative time in minutes | At procedure
  The difference in operative time (knife to skin - dressings on) and theatre time (into anaesthetic room - out of theatre) between the treatment arms will be compared.
Patient reported outcomes - Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 6 and 12 months post-surgery
  KOOS is a patient reported outcome measure derived from 5 subscales; symptoms (including stiffness), pain, function (daily living), function (sports and recreation activities) and quality of life with scores ranging from 0 - 100, a higher score indicating better health.
Patient reported outcomes - EQ-5D-5L (EuroQol, 5 Dimension, 5 Levels) | Baseline, 6 and 12 months post-surgery
  The EQ-5D-5L is a validated, generalised, health related quality of life questionnaire consisting of 5 domains related to daily activities with a 5-level answer possibility, which will be converted into multi-attributed utility scores using established algorithms.
Patient reported outcomes - Visual analogue scale (VAS) pain score | Baseline, 6 and 12 months post-surgery
  VAS will be used to measure patient reported pain. Patients will be requested to mark on a scale of 0 (no pain) to 10 (worst possible pain) the number that represents their knee pain. A second VAS score will measure soft tissue irritation. Patients will be requested to mark on a scale of 0 (no irritation) to 10 (worst possible irritation) the number that represents their amount of irritation they feel from the plate in their knee.
Patient reported outcomes - University of Carolina, Los Angeles Activity Score (UCLA Activity Score) | Baseline, 6 and 12 months post-surgery
  The UCLA Activity Score is a scale ranging from 1 to 10. The patient indicates their most appropriate activity level, with 1 defined as "wholly inactive, dependent on others, and cannot leave residence" and 10 defined as "regularly participates in impact sports".
Patient reported outcomes - Satisfaction and transition | 6 and 12 months post-surgery
  Participants will be asked how satisfied they are with their knee, how the problems related to their knee compare to before their operation and how willing they would be to have the operation again. General health will also be collected, and the participants will be asked to compare their general health now, to one year ago.
Patient reported outcomes - Health resource use (visits to primary care and hospital care services) | 6 and 12 months post-surgery
  This study will collect information on participants' health resource use, including time in operating theatre, visits to primary care, and hospital care services, during the follow-up. Summaries will be presented by trial arm and mean differences with 95% confidence intervals.
Knee range of motion (ROM) | 9 months post-randomisation (6 months post-surgery)
  ROM flexion and extension will be measured (in degrees) at baseline and nine months post randomisation.
Safety - rates of AEs / ADEs | Up to one year post-surgery
  Safety data will be collected throughout the duration of the trial, to determine the rates of Adverse Events and Adverse Device Effects.
Examine relationship between correction, change in loading and clinical outcomes (Calculated change in knee loading resulting from osteotomy correction from computer models of each patient). | 9 months post-randomisation (6 months post-surgery)
  Computer models based upon the CT geometry and informed by the achieved correction and video vector analysis will be used to calculate the change in knee loading due to the HTO surgery for each patient. This will enable the relationship between amount of correction, change in loading and outcome to be examined with the aim of optimising HTO surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Richie Gill, Prof, Principal Investigator — University of Bath
Locations (7):
- United Kingdom (7):
  - Royal United Hospitals NHS Trust, Bath, Avon
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Cardiff and Vale University Health Board, Cardiff, Wales
  - Royal Orthopaedic Hospital, Birmingham, West Midlands
  - Walsall Manor Hospital, Walsall, West Midlands
  - Great Western Hospital, Swindon, Wiltshire
  - Royal Devon and Exeter NHS Foundation Trust, Exeter

IPD SHARING:
Plan to Share IPD: No